CLINICAL TRIAL: NCT03037736
Title: Outpatient Performed Pterygium Surgery Study
Acronym: OPPS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding not received.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPPS
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Pterygium of Conjunctiva and Cornea
MeSH Terms: conditions — Pterygium Of Conjunctiva And Cornea | interventions — Fluorouracil; Bevacizumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: patients, physicians and evaluators will be masked as to the assignment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Patients will receive 0.1mL of normal saline injected subconjunctival in the area of the excised pterygium and 1 and 2 months postoperative.
  Interventions: Drug: Normal saline
- 5-Fluorouracil (Active Comparator): Patients will receive 0.1mL of 5-Fluorouracil, 5mg/0.1mL, injected subconjunctival in the area of the excised pterygium and 1 and 2 months postoperative.
  Interventions: Drug: 5-Fluorouracil
- Bevacizumab (Active Comparator): Patients will receive 0.1mL of bevacizumab, 2.5mg/0.1mL, injected subconjunctival in the area of the excised pterygium and 1 and 2 months postoperative.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: 5-Fluorouracil — 5-fluorouracil is an antimetabolite that is commonly used in glaucoma surgery to prevent postoperative scaring.
  Arms: 5-Fluorouracil
Drug: Bevacizumab — Bevacizumab is an anti-VEGF antibody that is commonly used to prevent or treat neovascularization in retinal disorders.
  Arms: Bevacizumab
Drug: Normal saline — Normal saline will be used as the placebo.
  Arms: Placebo

SUMMARY:
This is a randomized controlled trial of postoperative bevacizumab or 5-fluorouracil subconjunctival injections vs placebo for the recurrence of pterygia after excision using conjunctival autograft.

DETAILED DESCRIPTION:
Patients will be randomized at enrollment to one of three arms: 5-Fluorouracil (5-FU) 5mg/0.1mL, bevacizumab 2.5mg/0.1mL, or placebo. The placebo will be sterile, preservative-free injectable 0.9% normal saline. All patients will undergo pterygium excision surgery in the minor procedure room using a standardized surgical technique with conjunctival autograft. All patients will have a standardized postoperative drop protocol of neomycin/polymyxin/dexamethasone ointment four times daily for 2 weeks and fluorometholone drops 4 times daily for 2 weeks, three times daily for 2 weeks, twice daily for 2 weeks, once daily for 2 weeks then stopping.

At the 1-month and 2-month postoperative visits, patients will receive a subconjunctival injection based on their randomization assignment (5-FU, bevacizumab or placebo) in the area of the excised pterygium at least 1 mm posterior to the limbus. The total injected volume will be 0.1mL for all adjuvants.

The primary outcome will pterygium recurrence at 3 months, defined as evidence of at least 1 mm of fibrovascular growth onto the cornea. After the 3 month visit, patients who are determined to have a recurrence will be unmasked, and can received monthly 5-FU or bevacizumab injections at the discretion of the treating physician. Each of these visits will be treated as a study visit, and will be documented.

All patients will have study visits at the 6 and 12 month mark. If at any point any patient develops evidence of progression of recurrence, they may undergo further monthly 5-FU or bevacizumab injections at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic single-headed primary pterygia extending 2mm or more onto the cornea and determined by the physician to be a good candidate for surgical excision.
* Able to express a basic understanding of the study as determined by the treating physician.
* Age 18 and older.
* Commitment to return for follow up visits

Exclusion Criteria:

* Patients who are pregnant or who are planning on becoming pregnant during the study period
* Patients who are unable to tolerate subconjunctival injections in the clinic setting
* Patients with a diagnosis of glaucoma who are on more than 1 topical medication to control their intraocular pressure or who have ocular hypertension with a pressure of greater than or equal to 24mmHg.
* Patients with a previous history of conjunctival surgery in the eye with the pterygium
* Patients with a history of autoimmune or inflammatory conjunctival or corneal disorders, including but not limited to Stevens Johnson syndrome, graft versus host disease, mucous membrane pemphigoid, severe atopy, and herpes simplex epitheliitis or keratitis.
* Patients with an allergy to one or more of the study drugs.
* Patients who are on systemic immunosuppressive therapy or chemotherapy.
* Patients with a condition requiring topical steroid drops in the study eye or oral prednisone at a dose of more than 5mg/day.
* Patients with a history of scleritis or other severe ocular surface disease such as limbal stem cell deficiency.
* Patients with poor vision (defined as VA 20/200 or worse) in the contralateral eye.
* Patients with a large pterygium judged clinically to need amniotic membrane rather than a conjunctival autograft.
* Patients with bi-headed pterygia.
* Patients unable to undergo conjunctival autograft for any reason.
* Patients who are unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Recurrence | 3 months
  Recurrence of fibrovascular growth greater than or equal to 1mm onto cornea in area of excised pterygium as judged from slit lamp photographs by masked graders.

SECONDARY OUTCOMES:
Recurrence | 6 months
  Recurrence of fibrovascular growth greater than or equal to 1mm onto cornea in area of excised pterygium as judged from slit lamp photographs by masked graders.
Recurrence | 12 months
  Recurrence of fibrovascular growth greater than or equal to 1mm onto cornea in area of excised pterygium as judged from slit lamp photographs by masked graders.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Schallhorn, MD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: Undecided